CLINICAL TRIAL: NCT02572453
Title: Phase 2 Trial of the Heat Shock Protein-90 (Hsp90) Inhibitor AT13387 (Onalespib) in Patients With Relapsed/Refractory ALK+ ALCL, Mantle Cell Lymphoma, and BCL6+ DLBCL
Brief Title: Phase 2 Study of AT13387 (Onalespib) in ALK+ ALCL, MCL, and BCL-6+ DLBCL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug supply issues
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01681; NCI-2015-01681 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16-712; 9875 (Other: Dana-Farber - Harvard Cancer Center LAO); 9875 (Other: CTEP); UM1CA186690 (NIH); UM1CA186709 (NIH)
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Results first posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Recurrent Anaplastic Large Cell Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Transformed Non-Hodgkin Lymphoma; Refractory Anaplastic Large Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Transformed Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell | interventions — (2,4-dihydroxy-5-isopropylphenyl)-(5-(4-methylpiperazin-1-ylmethyl)-1,3-dihydroisoindol-2-yl)methanone

STUDY DESIGN:
Intervention Model Description: Patients are enrolled onto one of three parallel, non-comparative arms by disease type; treatment regimens are the same for each arm.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ALK+ ALCL (Experimental): Patients receive 160-mg/m2 onalespib by IV over 1 hour on days 1, 2, 8, 9, 15, and 16 of each 28-day cycle. Patients will continue on treatment indefinitely as long as they are responding and tolerating treatment.
  Interventions: Drug: Onalespib
- Relapsed MCL (Experimental): Patients receive 160-mg/m2 onalespib by IV over 1 hour on days 1, 2, 8, 9, 15, and 16 of each 28-day cycle. Patients will continue on treatment indefinitely as long as they are responding and tolerating treatment.
  Interventions: Drug: Onalespib
- BCL6+ DLBCL (Experimental): Patients receive 160-mg/m2 onalespib by IV over 1 hour on days 1, 2, 8, 9, 15, and 16 of each 28-day cycle. Patients will continue on treatment indefinitely as long as they are responding and tolerating treatment.
  Interventions: Drug: Onalespib

INTERVENTIONS:
Drug: Onalespib — Given IV
  Other Names: AT 13387; AT-13387; AT13387

SUMMARY:
This phase II trial studies how well onalespib works in treating patients with anaplastic large cell lymphoma, mantle cell lymphoma, or diffuse large B-cell lymphoma that has not responded to previous treatment (refractory) or that has returned after a period of improvement (recurrent). Onalespib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Overall response rate (ORR) to single agent AT13387 (onalespib) as measured by the proportion of partial and complete responses (PR + CR) in patients with relapsed/refractory ALK positive (+) anaplastic large cell lymphoma (ALCL), mantle cell lymphoma (MCL), and BCL6+ diffuse large B cell lymphoma (DLBCL).

SECONDARY OBJECTIVES:

I. Progression free survival (PFS) and overall survival (OS), as well as duration of response (DOR) of single agent AT13387 (onalespib) in patients with ALK+ ALCL, MCL, and BCL6+ DLBCL.

II. Safety and tolerability of single agent AT13387 (onalespib) in patients with ALK+ ALCL, MCL, and BCL6+ DLBCL.

EXPLORATORY OBJECTIVES:

I. Measurement of on-target activity of AT13387 (onalespib) in ALK+ ALCL, MCL, and BCL6+ DLBCL through immunoblotting and immunohistochemistry of pre-treatment, on-treatment, and time of progression tumor biopsies for HSP90 clients.

II. Determination of genetic and transcriptional markers for response and resistance to AT13387 (onalespib) in patients with ALK+ ALCL, MCL, and BCL6+ DLBCL.

OUTLINE:

Patients receive onalespib intravenously (IV) over 1 hour on days 1, 2, 8, 9, 15, and 16. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed, relapsed/refractory ALK+ ALCL (with ALK positivity defined by immunohistochemistry and/or fluorescence in situ hybridization [FISH]/cytogenetics from any prior biopsy), MCL, or BCL6+ DLBCL (with BCL6 positivity defined by immunohistochemistry from any prior biopsy) and meet the following criteria:
* Patients must have measurable disease that has not been previously irradiated, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional imaging or >= 10 mm with spiral computed tomography (CT) scan; if the patient has been previously irradiated, there must be evidence of progression since the radiation

  * Please note, this trial includes mandatory tumor biopsies pre-treatment, during cycle 1 and at the time of disease progression of accessible tumor; having accessible tumor for biopsy is not required for eligibility; we expect that at least 80% of patients will have accessible tumor for these biopsies, however
* Prior therapy

  * Please note, the washout period for prior therapies cannot be shortened
  * Please note, prior therapies can be from any time in the past
* ALK+ ALCL: patients must have disease that has relapsed and or is refractory to prior therapy, which must have included a multiagent chemotherapy regimen including an anthracycline, if not contraindicated, and prior brentuximab; prior crizotinib or other ALK inhibitor therapy, while recommended, is not mandatory; patients must have relapsed following or be ineligible for, or refuse, autologous stem cell transplant
* MCL: patients must have disease that has relapsed and or is refractory to prior therapy, which must have included a multiagent chemotherapy regimen and prior ibrutinib or other BTK inhibitor therapy; patients must have relapsed following or be ineligible for, or refuse, autologous stem cell transplant
* BCL6+ DLBCL: patients must have disease that has relapsed and or is refractory to prior therapy, which must have included an anthracycline, if not contraindicated; patients must have relapsed following or be ineligible for, or refuse, autologous stem cell transplant
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 75,000/mcL, unless due to marrow involvement by lymphoma in which case a platelet count of >= 30,000/mcL will be used
* Total bilirubin =< 1.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome or hemolysis, in which case =< 3.0 x ULN is allowed
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional upper limit of normal
* Creatinine =< 1.5 x ULN or a creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Potassium above the institutional lower limit of normal (supplementation to meet this is allowed)
* Magnesium above the institutional lower limit of normal (supplementation to meet this is allowed)
* Human immunodeficiency virus (HIV)+ patients are eligible for the trial provided they meet the other study criteria in addition to the following:

  * CD4+ T-cells >= 250/mm^3
  * HIV sensitive to antiretroviral therapy
  * Zidovudine not allowed
  * Long term survival anticipated on the basis of HIV alone were it not for the lymphoma
  * No concurrent acquired immunodeficiency syndrome (AIDS)-defining illness other than the lymphoma
* The effects of AT13387 (onalespib) on the developing human fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 months after the completion of AT13387 (onalespib) administration; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of AT13387 (onalespib) administration
* Although the pharmacokinetic (PK) data in humans is still unknown, the potential for drug-interaction cannot be ruled out; pre-clinical studies suggest that AT13387 (onalespib) is a substrate of P-glycoprotein (P-gp), a moderate inhibitor of BCRP and P-gp, and a strong inhibitor of MATE 1/2-K; patients must be willing to not take St. John wort or grapefruit juice while participating in this trial and should avoid drugs that are strong inducers of P-gp, and to switch to alternative drugs when available
* Hepatitis B positive patients are eligible; prophylactic hepatitis B virus (HBV) therapy is recommended but only if there is no circulating virus detectible
* Transformed lymphoma patients are eligible
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; steroids for symptom palliation are allowed, but must be either discontinued or on stable doses at the time of initiation of protocol therapy
* Patients who are receiving any other investigational agents; all investigational agents other than ibrutinib must have been discontinued at least 4 weeks prior to beginning treatment; prior ibrutinib therapy must have been discontinued at least 2 weeks prior to beginning therapy
* Patients with known leptomeningeal or brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; imaging or spinal fluid analysis to exclude central nervous system (CNS) involvement is not required, unless there is clinical suspicion by the treating investigator
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AT13387 (onalespib)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

  * There will be no exclusion of patients with known visual impairment or symptoms, including by not limited to peripheral flashes (photopsia), blurred or double vision, floaters, color distortion and dimness, difficulties with light/dark accommodation, tunnel vision or other field defects, halos, apparent movement of stationary objects, and complex disturbances; patients will have a baseline ophthalmologic exam to serve as a point of comparison and further exams as needed should visual symptoms develop; no pretreatment eye exam findings or ocular symptoms have been associated with an increased risk of ocular toxicity seen with AT13387
* Pregnant women are excluded from this study because AT13387 (onalespib) has the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AT13387 (onalespib), breastfeeding should be discontinued if the mother is treated with AT13387 (onalespib)
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Prior history of another malignancy (except for non-melanoma skin cancer or in situ cervical or breast cancer) unless disease free for at least three years; patients with prostate cancer are allowed if prostate specific antigen (PSA) is less than 1
* Patients should not receive immunization with attenuated live vaccine within one week of study entry or during study period
* History of noncompliance to medical regimens
* Consistent corrected QT (QTc) > 450 msec for men and > 470 msec for women by Fridericia formula, on 3 separate electrocardiograms (ECGs)
* Left ventricular ejection fraction (LVEF) < 50%, regardless of whether there are symptoms of heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caron A Jacobson, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (19):
- United States (19):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- ALK+ ALCL: Relapsed ALK+ ALCL, following Brentuximab and transplant ineligible (n=10 planned)
- Relapsed MCL: Relapsed MCL, following Ibrutinib and transplant ineligible (n=20 planned)
- BCL6+ DLBCL: Relapsed BCL6+ DLBCL, transplant ineligible (n=20 planned)
Period: Overall Study
Arm/Group | ALK+ ALCL | Relapsed MCL | BCL6+ DLBCL
Started | 1 | 4 | 20
Completed | 1 | 4 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALK+ ALCL | Relapsed MCL | BCL6+ DLBCL | Total
Number analyzed (Participants) | 1 | 4 | 20 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 12 | 15
  >=65 years | 0 | 2 | 8 | 10
Age, Continuous [Median (Full Range); unit: years] | 36 [36 to 36] | 66 [60 to 72] | 64 [25 to 84] | 64 [25 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 6 | 7
  Male | 1 | 3 | 14 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 4 | 17 | 22
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 1 | 4 | 17 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response (OR) = Complete + Partial (CR + PR)
  Per International Harmonization Project for lymphoma criteria, CR is defined as the disappearance of all evidence of disease. For FDG-avid or PET positive sites of disease prior to therapy, a mass of any size is permitted if PET negative; for variably FDG avid or PET negative lesions, regression to normal size on CT is necessary. The spleen or liver must also be nonpalpable with disappearance of any nodules, and the bone marrow, if initially involved, must be cleared on repeat biopsy.
  PR is defined as regression of measurable disease and no new sites of disease: a >50% decrease in the sum of the diameters of the up to 6 largest dominant masses with no increase in size of other masses. If the sites of disease were PET positive at baseline, there must be at least one previously involved site that remains PET positive.
Time Frame: Assessed every 2 cycles during treatment until disease progression; patients who discontinue for reasons other than progression will be evaluated every 6 months for up to 1 year after ending treatment or until progression or next therapy
Measure: Count of Participants; unit: Participants
Arm/Group | ALK+ ALCL | Relapsed MCL | BCL6+ DLBCL
Number analyzed (Participants) | 1 | 4 | 20
Participants | 0 | 0 | 2

2. Secondary Outcome: Frequency of Toxicities
Description: Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (version 5.0 is used staring April 1, 2018). Toxicities will be summarized with counts and proportions within each cohort and overall.
Time Frame: Assessed days 1, 2, 8, 9, 15, 16 of each 28-day cycle during treatment until progression; patients who discontinue for reasons other than progression evaluated every 6 months for up to 1 year after ending treatment or until progression or next therapy
Population: All patients who received any amount of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | ALK+ ALCL | Relapsed MCL | BCL6+ DLBCL
Number analyzed (Participants) | 1 | 4 | 20
Participants
  Any grade | 1 | 4 | 19
  Grade 1 (highest) | 1 | 1 | 1
  Grade 2 (highest) | 0 | 2 | 4
  Grade 3 (highest) | 0 | 0 | 7
  Grade 4 (highest) | 0 | 1 | 7

3. Secondary Outcome: Progression-free Survival
Description: The progression-free survival will be estimated by Kaplan-Meier method. Progressive disease is defined by the International Harmonization Project for lymphoma criteria: any new lesion or an increase by > 50% of previously involved sites from nadir. This includes the appearance of any new lesion(s) > 1.5cm in any axis, a > 50% increase in the sum of diameters of > 1 site of disease or > 50% increase in the longest diameter of a previously identified node >1cm in short axis. If the sites of disease were PET positive at baseline, they must remain PET positive.
Time Frame: From the date of study entry until documentation of first progression or death from any cause; progression assessed every 2 cycles during treatment until disease progression or death
Measure: Median (Full Range); unit: months
Arm/Group | ALK+ ALCL | Relapsed MCL | BCL6+ DLBCL
Number analyzed (Participants) | 1 | 4 | 20
months | 1.8 [1.8 to 1.8] | 2.0 [1.2 to 3.1] | 1.8 [0.4 to 8.8]

4. Secondary Outcome: Overall Survival
Description: The overall survival will be estimated by Kaplan-Meier method. Median follow-up time will be assessed using the reverse Kaplan-Meier method.
Time Frame: From the date of study entry until death from any cause; assessed every 6 months for up to 1 year after ending treatment
Measure: Median (Full Range); unit: months
Arm/Group | ALK+ ALCL | Relapsed MCL | BCL6+ DLBCL
Number analyzed (Participants) | 1 | 4 | 20
months | 1.6 [1.6 to 1.6] | 7.5 [1.1 to 7.5] | 2.9 [0.6 to 8.8]

5. Secondary Outcome: Duration of Response
Description: Duration of response will be evaluated only in patients who respond with either a partial response or complete response while on study.
Time Frame: From first objective response (partial response or complete response) until the first date of documented progression assessed every 2 cycles or death due to any cause; assessed every 6 months up to 1 year after ending treatment
Population: Patients who achieved partial or complete response, n=2 of 25
Measure: Median (Full Range); unit: months
Arm/Group | ALK+ ALCL | Relapsed MCL | BCL6+ DLBCL
Number analyzed (Participants) | 0 | 0 | 2
months |  |  | 6.1 [0.03 to 6.1]

6. Other Pre Specified Outcome: Change in Protein Levels of BCL6 in Diffuse Large B Cell Lymphoma
Description: Will be assessed via immunohistochemistry. Comparisons will be made between baseline, on treatment, and time of progression protein levels and changes will be characterized as differences and as differences at the referenced time point as a proportion of baseline levels. An H-score will be used. The Wilcoxon rank sum test will be used to compare changes between responders and non-responders and a one-sided significance level will be used.
Time Frame: Assessed days 1, 8, 15 of each 28-day cycle and at treatment completion visit
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Protein Levels of Cyclin D1 in Mantle Cell Lymphoma
Description: as for outcome 6
Time Frame: Assessed days 1, 8, 15 of each 28-day cycle and at treatment completion visit
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Protein Levels of ALK in ALK+ Anaplastic Large Cell Lymphoma
Description: Will be assessed via immunohistochemistry. Comparisons will be made between baseline, on treatment, and time of progression protein levels. An H-score will be used. Results at each time point and as changes as a proportion of baseline levels will be reported descriptively.
Time Frame: Assessed days 1, 8, 15 of each 28-day cycle and at treatment completion visit
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Onalespib Activity
Description: Will be measured by changes in protein levels via immunoblotting. Will use a one-sided significance level.
Time Frame: Assessed days 1, 8, 15 of each 28-day cycle and at treatment completion visit
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Genetic and Transcriptional Analysis for Markers of Response and Resistance
Description: Will be assessed via exome sequencing and ribonucleic acid sequencing. Absolute algorithm will be used to determine the cancer cell fraction.
Time Frame: Assessed days 1, 8, 15 of each 28-day cycle and at treatment completion visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed days 1, 2, 8, 9, 15, 16 of each 28-day cycle during treatment until progression; patients who discontinue for reasons other than progression evaluated every 6 months for up to 1 year after ending treatment or until progression or next therapy. Patients who discontinue due to unacceptable toxicity will be followed until resolution
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting up until March 31, 2018. Starting April 1, 2018, CTCAE version 5.0 will be utilized for AE reporting. CTCAE version 5.0 became available prior to April 1, 2018.
Arm/Group | ALK+ ALCL | Relapsed MCL | BCL6+ DLBCL
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/4 | 13/20
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/4 | 5/20
Other Adverse Events (participants affected / at risk) | 1/1 | 4/4 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALK+ ALCL (N=1) | Relapsed MCL (N=4) | BCL6+ DLBCL (N=20)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Neutropenia (Investigations) | 0 (0) | 0 (0) | 2 (3)
Thrombocytopenia (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALK+ ALCL (N=1) | Relapsed MCL (N=4) | BCL6+ DLBCL (N=20)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (16) | 13 (36)
Platelet count decreased (Investigations) | 0 (0) | 4 (8) | 12 (28)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 8 (19)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (3) | 9 (27)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 8 (18)
White blood cell decreased (Investigations) | 0 (0) | 2 (2) | 7 (21)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (13)
Fatigue (General disorders) | 0 (0) | 1 (2) | 6 (14)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (3) | 5 (6)
Blurred vision (Eye disorders) | 0 (0) | 2 (2) | 4 (6)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 4 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (8) | 3 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5)
Alkaline phosphatase increased (Investigations) | 0 (0) | 3 (4) | 1 (3)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (13)
Headache (Nervous system disorders) | 0 (0) | 1 (6) | 3 (11)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (4)
Anorexia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (4)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (7)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 2 (4)
Flashing lights (Eye disorders) | 0 (0) | 0 (0) | 2 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Belching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3)
Sore on tongue (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Visual changes (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Weird dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT02572453/Prot_SAP_000.pdf